CLINICAL TRIAL: NCT01209520
Title: Pilot Study Targeting Residual Hypermethylation in Early Stage Non-Small Cell Lung Cancer As Part of Adjuvant Therapy and Preventive Strategy
Brief Title: Residual Hypermethylation in Early Stage Non-Small Cell Lung Cancer (NSCLC) As Part of Adjuvant Therapy and Preventive Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ikechukwu Akunyili, Assistant Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080779; SCCC-2008045 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2010-09-22; First posted 2010-09-27 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Lung Cancer; Non Small Cell Lung Carcinoma; Hypermethylation
Keywords: Lung Cancer; Non-Small Cell Lung Carcinoma; NSCLC; Methylation Analysis; Hypermethylation; Targeted Genes; Tumorigenesis; Tumor Supressor Genes
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinogenesis | interventions — Cisplatin; Carboplatin; Paclitaxel; Azacitidine; Blood Specimen Collection; Vinorelbine; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adjuvant Chemotherapy + Vidaza (Experimental)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Vidaza; Procedure: Tumor Specimen for Methylation Analysis; Procedure: Blood Sample for Methylation Analysis; Drug: Vinorelbine; Drug: Docetaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Cisplatin — Patients will receive a total of 4 cycles of adjuvant chemotherapy (each cycle given every 21 days). Conventional chemotherapy will be selected at discretion of the treating physicians except on those cases in which pathologic diagnosis indicates non squamous NSCLC.
  Other Names: Platinol®,; cis-diamminedichloroplatinum
Drug: Carboplatin — Patients will receive a total of 4 cycles of adjuvant chemotherapy (each cycle given every 21 days). Conventional chemotherapy will be selected at discretion of the treating physicians except on those cases in which pathologic diagnosis indicates non squamous NSCLC.
  Other Names: Paraplatin®
Drug: Paclitaxel — Patients will receive a total of 4 cycles of adjuvant chemotherapy (each cycle given every 21 days). Conventional chemotherapy will be selected at discretion of the treating physicians except on those cases in which pathologic diagnosis indicates non squamous NSCLC.
  Other Names: Taxol
Drug: Vidaza — Patient will receive 5-azacitidine at a dose of 75 mg/m2 intravenously daily on day 1-5 every 28 days for 6 cycles
  Other Names: 5-azacitidine
Procedure: Tumor Specimen for Methylation Analysis — Obtained from tissue of resected NSCLC tumor.
Procedure: Blood Sample for Methylation Analysis — Pre-Surgery, Post-Surgery, Post-Vidaza Therapy and during follow-up.
Drug: Vinorelbine — Patients will receive a total of 4 cycles of adjuvant chemotherapy (each cycle given every 21 days). Conventional chemotherapy will be selected at discretion of the treating physicians except on those cases in which pathologic diagnosis indicates non squamous NSCLC.
  Other Names: Navelbine®
Drug: Docetaxel — Patients will receive a total of 4 cycles of adjuvant chemotherapy (each cycle given every 21 days). Conventional chemotherapy will be selected at discretion of the treating physicians except on those cases in which pathologic diagnosis indicates non squamous NSCLC.
Drug: Pemetrexed — Patients will receive a total of 4 cycles of adjuvant chemotherapy (each cycle given every 21 days). Conventional chemotherapy will be selected at discretion of the treating physicians except on those cases in which pathologic diagnosis indicates non squamous NSCLC.

SUMMARY:
The trial investigates the feasibility and efficacy of targeting Non-Small Cell Lung Cancer (NSCLC) "driven" by epigenetic changes. The investigators study the impact of 5-azacitidine (Vidaza®, Celgene, Summit, NJ, USA) in combination with conventional cytotoxic chemotherapy in a sequential fashion. The study population consists of all NSCLC patients who undergo "curative" lung cancer resection and whose tumors harbor hypermethylation in any of the protocol-specific genes (samples will be banked for additional molecular testing including other 21 loci which have shown to be important in lung carcinogenesis.

DETAILED DESCRIPTION:
Adjuvant chemotherapy has become an essential part for the treatment of stage IB-IIIA NSCLC patients based on 4 randomized clinical trials showing survival advantage for patients who received adjuvant CT, oncologists initially started to adapt this modality of treatment for pathologically stage IB-IIIA NSCLC patients [4]. Herein, NSCLC patients will be treated in the adjuvant setting with conventional doublet platinum-based chemotherapy followed by 5-azacitidine, a demethylating agent. The planned dosages to be used in this trial have been extensively studied in previously conducted clinical trials involving all therapeutic agents.

All patients will undergo thorough surgical resection of the primary lung tumor, and evidence of promoter hypermethylation of gene(s) must be present in the tumor specimen and/or blood sample (plasma or WBC). The collection of tumor specimen will be considered a priority to correlate the tumor "methylation pattern/profile" with the serum "methylation pattern/profile". If tumor specimen is not available for any reason, but the patient has at least one of the 9 targeted genes hypermethylated in the serum, the patient is eligible to be enrolled into the trial.

Treatment will consist of 2 parts:

Part A. Adjuvant chemotherapy.

Following surgical resection of NSCLC and test positive for promoter hypermethylation in at least one (1) of the targeted TSGs described, patient will start adjuvant conventional chemotherapy (doublet platinum-based chemotherapy) for stage IB-IIIA NSCLC. In the case a patient with stage IB refuses adjuvant chemotherapy, the patient still can be enrolled into Part B of the study if he/she understands the concept of the trial and sign an informed consent.

Conventional chemotherapy will be selected at discretion of the treating physicians except on those cases in which pathologic diagnosis indicates non squamous NSCLC. Those patients will be treated with pemetrexed. Patients will receive a total of 4 cycles of adjuvant chemotherapy (each cycle given every 21 days). Pegfilgrastim, a granulocyte-colony stimulating factor (G-CSF), will be allowed on day 2 at discretion of the clinician.

All patients should be premedicated prior to paclitaxel or docetaxel administration in order to prevent severe hypersensitivity reactions (HSR). Such premedication may consist of: dexamethasone 20 mg orally administered approximately 12 and 6 hours before paclitaxel or docetaxel; diphenhydramine 50 mg intravenously and cimetidine (300 mg) or ranitidine (50 mg) intravenously 30 minutes before paclitaxel. In case of pemetrexed, patient will received an injection of vitamin B-12 1,000 mcg IM a week prior to start therapy as well as folic acid 1 mg po daily a week before pemetrexed infusion and during the entire course of treatment with this antifolate agent.

The dosages and toxicities of these chemotherapy agents are very well described in the clinical setting, and patients will be managed as any other patient receiving standard chemotherapy.

Part B. Targeted therapy using 5-azacitidine.

If the patient decides not to receive adjuvant chemotherapy, the patient still can be enrolled into the study, if the patient understands the concept of chemoprevention and consents to blood sampling during 5-azacitidine administration and follow-up (informed consent signed). This part of the study consists of 6 cycles of 5-azacitidine (Vidaza®, Celgene, Summit, NJ, USA).

Four weeks after completion of adjuvant chemotherapy (day 28 from day 1 of last cycle of chemotherapy), the patient will continue his/her treatment plan with 6 cycles of 5-azacitidine. To be eligible for this part of the study, patient must have no evidence of disease (NED). Thus, patient will be assessed by CT scan chest/abdomen/pelvis with and without intravenous contrast prior to initiating Part B. In case of iodine allergy/anaphylaxis history, patient will be assessed with MRI. Progression of disease will be defined by RECIST criteria.

Patient will receive 5-azacitidine at a dose of 75 mg/m2 intravenously daily on day 1-5 every 28 days for 6 cycles. Biological correlatives will be performed during this period. Toxicity management is described in section 6.0. The use of growth factor support (either erythropoietin stimulating agents or G-CSF) will be also allowed at discretion of the treating physician.

Anatomical Studies:

All patients will have surgical resection of the primary tumor. Pieces of the resected tumor and non-tumor lung tissues that are not required for pathological evaluation will be frozen in optimum temperature compound (OTC) and saved for molecular analysis.

As part of the enrollment process, patient will be assessed through CT scan of the chest/abdomen/pelvis with and without intravenous contrast or with MRI in case of contraindication for iodine contrast, prior to initiate Part B of the treatment (confirming clinically and radiological "no evidence of disease-NED"). Another assessment will be performed 4 weeks after the last dose of 5-azacitidine (to confirm NED status). Patient will be clinically followed up every 3 months until completion of 2 years post-treatment. Imaging tests will be performed every 3 months with CT scan as part of the standard follow-up until completion of 2 years post-surgery. After 2 years of post-treatment completion, patient will be followed up every 6 months in the clinic and also by radiographic studies until completion of 5 years post-treatment. In the case of clinical suspicion for progression, patient will undergo a thorough and complete work-up to rule out this possibility. This may include imaging diagnostic tests, biopsy, or other tests and procedures.

Biological Correlatives:

The premise of the study is that certain loci will be hypermethylated in the lung cancer specimen of the patients. For some loci (which we shall call Type I) the tumor will show significantly elevated methylation compared to adjacent histologically normal tissue, thus providing a cancer-specific methylation signal. Other loci (which we will refer to as Type II) may be methylated in the tumor as well as in the adjacent "histologically" normal tissue and/or WBCs. These loci will not be cancer-specific markers, though they may indicate precancerous changes or they may be indicative of "cancer risk". Their hypermethylation may be age-associated or environmentally induced, yielding "field effects" or "field defects". Field defects would consist of molecular alterations (in this case hypermethylation) that are not yet visible as histological changes.

Independent of whether a hypermethylated locus is specific for overt cancer (Type I) or not (Type II), it would be of interest for the study. These Type II changes would be "hypothesis generating". Since it has been well documented in the literature that DNA from cells can be shed into the blood stream (more so in the case of cancer patients), it would be expected that at least for some of the loci that are hypermethylated (Type I and II), this methylation would be detectable in the plasma. Tumor tissue methylation will be correlated with serum obtained at the time of tumor resection.

It might be expected that complete resection would lead to a reduction or complete disappearance in the methylation signal for Type I loci in the plasma, since the source of the signal has been removed. Type II also shows methylation in the tissue adjacent to the tumor, these loci might continue to provide signal in the plasma (though it may be somewhat diminished).

Type I loci would therefore be of great use to verify complete resection and to monitor recurrence (one would anticipate the signal to increase again as the cancer grows back), while Type II loci would be a great tool to monitor the efficacy of demethylating drugs. It must be acknowledged that the spectrum of Type I and Type II methylation may not be sharply delineated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologic diagnosis of NSCLC.
* Patients must have surgical resection for NSCLC (stage I-IIIA) and tumor specimen (ideally) and/or blood sample available for biological correlative studies.
* Patient's tumor specimen and/or blood sample must show hypermethylation in at least one (1) of the following genes: DAPK, RASSF1A, CDKN2A (p16INK4a), GATA-4, GATA-5, SPARC, MGMT, APC, and hMLH1.
* Patient's age must be 18 years or greater.
* Patients must have adequate organ and marrow function prior to be enrolled into the trial, as defined below:

  * Absolute neutrophil count (ANC) > 1500/mm3
  * Platelets > 100,000/mm3
  * Hemoglobin > 8.0 g/dL (with packed red blood cell transfusion or use of erythropoietin stimulating agents allowed)
  * Serum creatinine < 2.0 mg/dl.
  * Total bilirubin < 2.0 mg/dl.
  * AST/ALT < 2 x the upper limits of institutional normal.
* ECOG performance status of 0, 1, or 2.
* Estimated survival of > 12 months.
* Patients must be able to understand and agree to sign an IRB-approved informed consent form, including permission to draw blood sample for correlative studies during active treatment and follow-up.
* Women of child-bearing potential and men must agree to use adequate contraceptive method (hormonal or barrier method of birth control) prior to study entry for the duration of study.
* Women of childbearing potential must have a negative serum pregnancy test prior to start targeted therapy with 5-azacitidine.
* Patients with HIV infection (but not AIDS) are eligible for this trial. Therefore, no HIV testing will be required.

Exclusion Criteria:

* Patients who are not candidates for surgical resection.
* Patients who have received radiation therapy.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, breast DCIS adequately treated, or other cancer for which the subject has been disease-free ≥ 5 years.
* Subjects should not have a significant history of cardiac disease (e.g., unstable angina, congestive heart failure, or uncontrolled arrhythmias).
* Subjects must not have an uncontrolled seizure disorder, or active neurological disease.
* Patients who have significant systemic infections including AIDS.
* Pregnant and/or lactating women.
* Known or suspected hypersensitivity to azacitidine or mannitol.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ikechukwu Akunyili, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjuvant Chemotherapy + Vidaza
Started | 6
Completed | 3
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adjuvant Chemotherapy + Vidaza
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 74.5 [61 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Showing a Presence of Methylated Tumor Suppressor Genes in Their Tumor Tissue and/or Serum Achieving Partial or Complete Response to Protocol Therapy.
Description: To determine the feasibility and efficacy of incorporating a demethylating agent (5-azacitidine; Vidaza®, Celgene, Summit, NJ, USA) as part of adjuvant therapy in patients diagnosed with NSCLC who harbor methylated tumor supressor genes (TSGs) in their tumor tissue and/or serum. Response to be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.0.
Time Frame: Up to 2 years
Population: Study data were not analyzed due to insufficient number of evaluable patients.
Arm/Group | Adjuvant Chemotherapy + Vidaza
Number analyzed (Participants) | 0

2. Primary Outcome: Degree of Demethylation in Patient Tumor Tissue and/or Serum Induced by 5-azacitidine on Specific Tumor Specific Genes (TSGs)
Description: To measure the grade of demethylation induced by 5-azaciditine on specific TSGs by analyzing plasma DNA, and global demethylation by analyzing WBC DNA, and determine the duration of this effect.
Time Frame: Up to 2 years
Population: Study data were not analyzed due to insufficient number of evaluable patients.
Arm/Group | Adjuvant Chemotherapy + Vidaza
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Adjuvant Chemotherapy + Vidaza
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Chemotherapy + Vidaza (N=6)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Chemotherapy + Vidaza (N=6)
Abdominal Pain (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Bone pain (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Metabolism and nutrition disorders) | 1 (5)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dermatology - Skin, other (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema - limbs (Blood and lymphatic system disorders) | 1 (1)
Edema - head and neck (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 2 (4)
Hemolysis (Blood and lymphatic system disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Joint pain (General disorders) | 1 (2)
Large intestinal mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Neurology - other (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Petechiae (Blood and lymphatic system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Taste alteration (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis/thrombus/embolism (Blood and lymphatic system disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study data were not analyzed due to insufficient number of evaluable patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes